CLINICAL TRIAL: NCT02933528
Title: An Open-Label, Safety Study to Assess the Potential for Adrenal Suppression Following Maximal Use Treatment With DSXS in Patients With Moderate to Severe Scalp Psoriasis
Brief Title: Safety Study to Assess the Potential for Adrenal Suppression Following Maximal Use Treatment With DSXS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSXS 1538a
Record Dates: First submitted 2016-10-11; First posted 2016-10-14 (Estimated); Results first posted 2018-12-06 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-11

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dsxs topical product (Experimental): treatment with DSXS once daily for 28 days
  Interventions: Drug: DSXS Topical product

INTERVENTIONS:
Drug: DSXS Topical product — once daily for 28 days
  Other Names: Active

SUMMARY:
An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Maximal Use Treatment with DSXS .

DETAILED DESCRIPTION:
Evaluate the potential of DSXS topical product to suppress HPA axis function in patients with moderate to severe scalp psoriasis. Evaluate the efficacy parameters and adverse event (AE) profiles of DSXS topical product administered to patients with moderate to severe scalp psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating females 18 years of age or older.
* IRE-approved, signed informed consent form that meets all criteria of current FDA regulations.

Exclusion Criteria:

* Females who are pregnant, nursing, planning to become pregnant during the duration of the study, or if of child-bearing potential and sexually active and not prepared to use appropriate contraceptive methods to avoid pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-07-11 (Actual); Primary Completion 2017-08-11 (Actual); Study Completion 2017-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novum Pharmaceutical Research Services, Study Chair — http://www.novumprs.com/contact
Locations (1):
- Taro Pharmaceuticals USA, Inc., Hawthorne, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dsxs Topical Product
Started | 24
Completed | 22
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Dsxs Topical Product
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (17.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 3
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Percent Scalp Affected with Plaque Psoriasis [Mean (Standard Deviation); unit: percent of scalp] | 42.2 (22.6)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients in the Study With HPA Axis Suppression
Description: Hypothalamic Pituitary Adrenal (HPA) Axis Response to stimulation
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Dsxs Topical Product
Number analyzed (Participants) | 14
Participants
  Yes | 1
  No | 13

ADVERSE EVENTS:
Time Frame: 1 year, 1 month
Arm/Group | Dsxs Topical Product
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 1/23
Other Adverse Events (participants affected / at risk) | 6/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dsxs Topical Product (N=23)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dsxs Topical Product (N=23)
Conjunctival haemorrhage (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Application site alopecia (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Chemical burn of skin (Injury, poisoning and procedural complications) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Sinus headache (Nervous system disorders) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-12-27): https://cdn.clinicaltrials.gov/large-docs/28/NCT02933528/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-18): https://cdn.clinicaltrials.gov/large-docs/28/NCT02933528/SAP_001.pdf